CLINICAL TRIAL: NCT02890979
Title: Next Generation Sequencing of Esophageal Cytology for the Early Detection of Esophageal Cancer
Brief Title: Swallowable Sponge Cell Sampling Device and Next Generation Sequencing in Detecting Esophageal Cancer in Patients With Low or High Grade Dysplasia, Barrett Esophagus, or Gastroesophageal Reflux Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00015499; NCI-2016-01318 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00015499 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Barrett Esophagus; Dysplasia; Esophageal Adenocarcinoma; Esophageal Squamous Cell Carcinoma; Gastroesophageal Reflux Disease; Metaplasia
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma; Gastroesophageal Reflux; Metaplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (1):
- Screening (cytology collection) (Experimental): Patients undergo cytology specimen collection procedure using a swallowable sponge cell sampling device.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Device: Swallowable Sponge Cell Sampling Device

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Undergo cytology specimen collection procedure using a swallowable sponge cell sampling device
  Other Names: Cytologic Sampling
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Device: Swallowable Sponge Cell Sampling Device — Undergo cytology specimen collection procedure using a swallowable sponge cell sampling device
  Other Names: Swallowable Sponge; Swallowable Sponge Device

SUMMARY:
This pilot clinical trial studies how well a swallowable sponge cell sampling device and next generation sequencing work in detecting esophageal cancer in patients with low or high grade dysplasia, Barrett esophagus, or gastroesophageal reflux disease. Checking biomarkers in abnormal esophageal cells using a swallowable sponge cell sampling device and next generation sequencing may improve diagnosis and treatment of esophageal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the sensitivity and specificity of next generation sequencing for the detection of esophageal cancer from esophageal sponge cytology specimens.

SECONDARY OBJECTIVES:

I. Determine the ability of next generation gene sequencing (NGS) of esophageal sponge samples to collect an adequate sample to detect mutations that are present in the underlying tissue.

II. Determine the cost associated with esophageal cytology with next generation genome sequencing as a screening tool.

III. Continue to collect safety and tolerability data related to the use of the Oesotest esophageal sponge.

IV. Determine the limitations of esophageal sponge cytology and future needs to improve this technique.

V. Use the data collected to design a larger screening trial to determine the ability of esophageal cytology with next generation sequencing to screen for esophageal cancer in the general population.

OUTLINE:

Patients undergo cytology specimen collection procedure using a swallowable sponge cell sampling device.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Patients must be scheduled for a procedure capable of providing a definitive pathologic diagnosis and evaluating for complications of the esophageal sponge on the same day as the study procedure, either upper endoscopy or surgical esophagectomy
* One of the following inclusion criteria must be true for patient to be eligible for enrollment:
* Subjects with known esophageal cancer (adenocarcinoma or squamous cell carcinoma)
* Subjects with a history of low or high grade dysplasia
* Subjects with risk factors for esophageal malignancy including Barrett?s esophagus and gastroesophageal reflux disease (GERD)

Exclusion Criteria:

* Subjects that are unable to swallow a tablet/pill
* Subjects with completely obstructing esophageal cancer
* Subjects with known or suspected esophageal varices
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Any condition which, in the opinion of the investigator precludes the patient from completion of the study procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-08-03 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Detection of gene mutations using next generation sequencing (NGS) | Up to 2 years
  Will calculate the concordance of the gene mutations identified from the sponge sample to those identified from the tissue biopsy (control).

SECONDARY OUTCOMES:
Sensitivity and specificity of the NGS probes to detect underlying esophageal dysplasia or cancer | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: James Dolan, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States